CLINICAL TRIAL: NCT03558750
Title: Combination of Rituximab, Lenalidomide and Nivolumab for Relapsed/ Refractory Non-germinal Center (Non-GCB) Type Diffuse Large B Cell Lymphoma (DLBCL) Including Primary Central Nervous System Lymphoma (PCNSL): A Phase 1/2 Trial
Brief Title: Rituximab, Lenalidomide, and Nivolumab in Treating Participants With Relapsed or Refractory Non-Germinal Center Type Diffuse Large B Cell Lymphoma or Primary Central Nervous System Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Nishitha Reddy, MD, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC PCL 1758; NCI-2018-01092 (Registry Identifier: NCI, Clinical Trials Reporting Program)
Record Dates: First submitted 2018-06-04; First posted 2018-06-15 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Recurrent Central Nervous System Lymphoma; Recurrent Diffuse Large B-Cell Lymphoma; Refractory Central Nervous System Lymphoma; Refractory Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Nivolumab; Rituximab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (nivolumab, rituximab, lenalidomide) (Experimental): Nivolumab give by IV over 60 minutes on days 1 and 15, rituximab IV on day 1, and lenalidomide by mouth once per day on days 1-21. Repeats every 28 days for up to of 8 courses in the absence of disease progression or unacceptable toxicity. Patients with partial response or stable disease at the end of 8 cycles will be offered lenalidomide and nivolumab maintenance for up to 12 courses.
  Interventions: Biological: Nivolumab; Biological: Rituximab; Drug: Lenalidomide

INTERVENTIONS:
Biological: Nivolumab — Given by IV
Biological: Rituximab — Given by IV
Drug: Lenalidomide — Given by mouth

SUMMARY:
This phase I/II trial studies the side effects and best dose of lenalidomide when given in combination with rituximab and nivolumab and how well they work in treating participants with non-germinal center type diffuse large B cell lymphoma or primary central nervous system lymphoma that has come back or isn't responding to treatment. Monoclonal antibodies, such as rituximab and nivolumab, may interfere with ability of cancer cells to grow and spread. Drugs used in chemotherapy, such as lenalidomide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving rituximab, lenalidomide, and nivolumab may work better in treating participants with diffuse large B cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose and toxicity profile of lenalidomide in combination with standard doses of rituximab and nivolumab in relapsed/refractory (R/R) diffuse large B cell lymphoma (DLBCL) (non-germinal center B cell [non-GCB]) and in primary central nervous system (CNS) lymphoma (PCNSL) (Phase I).

II. Evaluate the efficacy of lenalidomide in combination with standard doses of rituximab and nivolumab in R/R non-GCB type DLBCL and PCNSL (Phase II).

SECONDARY OBJECTIVES:

I. To assess the safety and tolerability of nivolumab when combined with lenalidomide and rituximab.

II. To determine the time to progression (complete response, partial response or stable disease), progression free survival (PFS) and overall survival (OS).

III. To evaluate the difference in overall response rate between those with and without programmed cell death ligand 1 (PD-L1) protein expression in tumor (subgroup analysis).

IV. To evaluate the difference in overall response rate between those with and without MYD88 mutation in tumor (subgroup analysis).

EXPLORATORY OBJECTIVES:

I. To perform PD-L1, PD-1 expression on tumor cells by immunohistochemistry including double staining for PAX-5 and PD-L1 and CD68 and PD-L1, CD3/CD4/CD8 for T cell infiltration, CD68 for tumor associated macrophages.

II. To assess for presence of MYD88 L265 mutation by allele specific polymerase chain reaction (PCR) in tumor tissue and /or cerebrospinal fluid (CSF) (where lumbar puncture is clinically performed).

III. To perform fluorescence in situ hybridization (FISH) for 9p24.1/ PD-L1/PD-L2 locus.

IV. To evaluate MYD88 PCR on CSF (where available). V. To perform gene expression panel for tumor immune response in tumor samples (prioritizing cases in which a second serial biopsy is available).

OUTLINE: This is a phase I, dose-escalation study of lenalidomide followed by a phase II study.

Participants receive nivolumab intravenously (IV) over 60 minutes on days 1 and 15, rituximab IV on day 1, and lenalidomide orally (PO) once daily (QD) on days 1-21. Treatment repeats every 28 days for up to of 8 courses in the absence of disease progression or unacceptable toxicity. Patients with partial response (PR) or stable disease at the end of 8 cycles will be offered lenalidomide and nivolumab maintenance for up to 12 courses.

After completion of study treatment, participants are followed up every 3 months for 2 years and then every 6 months until year 4.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form.
* Able to adhere to the study visit schedule and other protocol requirements in the opinion of the investigator
* Patients with histological confirmation of relapsed/refractory non-GCB type (using Hans algorithm) diffuse large B cell lymphoma (DLBCL) or relapsed/refractory primary CNS lymphoma (PCNSL) with at least one of the following characteristics:

  * Definition of refractory disease: progression of disease based on Cheson criteria for DLBCL or international primary CNS lymphoma cooperative group for PCNSL either with nonresponse or progression within 3 months of prior therapy
  * Definition of relapsed disease: progression of disease based on Cheson criteria for DLBCL or International primary CNS lymphoma cooperative group for PCNSL at least 3 months after prior therapy
  * Definition of non-GCB subtype (Hans algorithm): cases will be subclassified based on immunohistochemical staining with CD10, BCL-6 and MUM-1 as previously described.
  * Patients should have exhausted (or be ineligible for) approved therapies known to provide clinical benefit for DLBCL or PCNSL (e.g. high dose chemotherapy with autologous stem cell transplant, chimeric antigen receptor-transduced [CAR-T] therapy, etc.).
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 2 at study entry.
* Absolute neutrophil count >= 1000/mm^3 within 45 days prior to initiation of therapy. (Patients with documented marrow involvement (with lymphoma) or hypersplenism secondary to involvement of the spleen by lymphoma at the time of randomization are not required to meet the parameter).
* Platelet count >= 75K /mm^3 within 45 days prior to initiation of therapy. (Patients with documented marrow involvement (with lymphoma) or hypersplenism secondary to involvement of the spleen by lymphoma at the time of randomization are not required to meet the parameter).
* Serum creatinine =< 2.0 mg/dL or creatinine clearance of > 40 ml/min within 45 days prior to initiation of therapy. (Patients with documented marrow involvement (with lymphoma) or hypersplenism secondary to involvement of the spleen by lymphoma at the time of randomization are not required to meet the parameter).
* Total bilirubin =< 1.5 mg/dL within 45 days prior to initiation of therapy. (Patients with documented marrow involvement (with lymphoma) or hypersplenism secondary to involvement of the spleen by lymphoma at the time of randomization are not required to meet the parameter).
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2 x upper limit of normal (ULN) within 45 days prior to initiation of therapy. (Patients with documented marrow involvement (with lymphoma) or hypersplenism secondary to involvement of the spleen by lymphoma at the time of randomization are not required to meet the parameter).
* Disease free of prior malignancies for >= 3 years with exception of currently treated basal cell or squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast.
* All study participants must be registered into the mandatory Revlimid Risk Evaluation and Mitigation Strategies (REMS) program, and be willing and able to comply with the requirements of the Revlimid REMS program. program, and be willing and able to comply with the requirements of the Revlimid REMS program.

  * Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10-14 days and again within 24 hours prior to prescribing lenalidomide for cycle 1 (prescriptions must be filled within 7 days as required by the Revlimid REMS program) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy.

  ** A female of childbearing potential is a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
* Able to take aspirin (81 or 325 mg) daily or for thromboprophylaxis with lenalidomide.

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent.
* Pregnant or breast feeding females (lactating females must agree not to breast feed while taking lenalidomide).
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Use of any other experimental drug or therapy within 28 days of baseline.
* Known hypersensitivity to thalidomide.
* Known prior development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Concurrent use of other anti-cancer agents or treatments.
* Patients with a prior history of pulmonary toxicity due to medications (Ex: history of carmustine [BCNU] toxicity).
* Active human immunodeficiency virus (HIV) infection or infectious hepatitis, type B or C.

  * Patients with a past or resolved hepatitis B virus (HBV) infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of hepatitis B surface antigen [HBsAg]) may be included if HBV deoxyribonucleic acid (DNA) is undetectable. If enrolled, patients must be willing to undergo monthly HBV DNA testing.
  * HIV positive patients may enroll if they meet all of the below criteria:

    * HIV is sensitive to antiretroviral therapy.
    * Must be willing to take effective antiretroviral therapy if indicated.
    * No history of CD4 prior to or at the time of lymphoma diagnosis < 300 cells/mm^3.
    * No history of acquired immunodeficiency syndrome (AIDS)-defining conditions.
    * If on antiretroviral therapy, must not be taking zidovudine or stavudine.
    * Must be willing to take prophylaxis for pneumocystis jiroveci pneumonia (PCP) during therapy and until at least 2 months following the completion of therapy or until the CD4 cells recover to over 250 cells/mm^3, whichever occurs later.
* A diagnosis of deep vein thromboses in the preceding four weeks of study enrollment.
* Subjects with active interstitial pneumonitis.
* Patient with active, uncontrolled infections (patients must be afebrile for > 48 hours off antibiotics).
* Patient with clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis.
* Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results or that could increase risk to the patient, including renal disease that would preclude chemotherapy administration or pulmonary disease (including obstructive pulmonary disease and history of bronchospasm).
* Major surgery within 4 weeks prior to cycle 1, other than for diagnosis.
* Malabsorption syndrome or other condition that precludes oral route of administration of lenalidomide.
* Vaccinations with a live vaccine within 28 days prior to start of treatment or need for live vaccine at any time during study treatment.
* Patient must not have serious medical or psychiatric illness likely to interfere with participation in this clinical study in the opinion of the investigator.
* Inability to swallow oral medications.
* Subjects with New York Heart Association (NYHA) class III or IV heart failure.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2019-04-16 (Actual); Study Completion 2019-04-16 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) (Phase I) | At the end of cycle 2 (each cycle is 28 days)
  The maximum-tolerated dose (MTD) is the highest dose at which no more than one dose limiting toxicities are observed among 6 subjects. The MTD of lenalidomide in combination with standard doses of rituximab and nivolumab will be determined from 3+3 design.
Overall response rate (complete response, partial response, or stable disease) (Phase II) | At the end of cycle 8 (each cycle is 28 days)
  Parametric tests such as t-test or the non-parametric statistical methods such as Wilcoxon rank sum will be used to compare differences in the means for endpoints of interest between response and non-response groups.

SECONDARY OUTCOMES:
Time to progression (complete response, partial response, or stable disease) | Up to 4 years
  Parametric tests such as t-test or the non-parametric statistical methods such as Wilcoxon rank sum will be used to compare differences in the means for endpoints of interest between response and non-response groups.
Progression free survival | From the time of enrollment in the study until progression, relapse, or death, assessed up to 4 years
  Survival curves will be calculated from the Kaplan-Meier method. The median PFS with 95% confidence will be reported. Cox regression will be applied to assess the association between PFS/OS.
Overall survival | From the time of enrollment in the study until death, assessed up to 4 years
  Survival curves will be calculated from the Kaplan-Meier method. The median OS with 95% confidence will be reported. Cox regression will be applied to assess the association between progression free survival/overall survival
Incidence of adverse events per national Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 4.03 | Up to 30 days after treatment
  Data from all subjects who receive any protocol therapy will be included in the safety analyses.
Difference in overall response rate between those with and without programmed cell death ligand 1 (PD-L1) protein expression in tumor (subgroup analysis) | Up to 4 years
  Parametric tests such as t-test or the non-parametric statistical methods such as Wilcoxon rank sum will be used to compare differences in the means for endpoints of interest between response and non-response groups.
Difference in overall response rate between those with and without MYD88 mutation in tumor (subgroup analysis) | Up to 4 years
  Parametric tests such as t-test or the non-parametric statistical methods such as Wilcoxon rank sum will be used to compare differences in the means for endpoints of interest between response and non-response groups.

CONTACTS AND LOCATIONS:
Overall Officials: Nishitha Reddy, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided